CLINICAL TRIAL: NCT07393880
Title: Non-Invasively Re-Training the Tinnitus Brain Using Bimodal Electrical-Sound Stimulation (NITESGON-ADT): Protocol for a Prospective, Double-Blind, Randomised Controlled Trial
Brief Title: Bimodal Electrical-Sound Stimulation and Auditory Training for Chronic Tonal Tinnitus
Acronym: NITESGON-ADT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dublin, Trinity College (Other)
Responsible Party: Principal Investigator, Sven Vanneste, Professor, University of Dublin, Trinity College
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: NITESGON-SPREC102020-46; DRG2332 (Other Grant/Funding Number: RNID)
Record Dates: First submitted 2026-01-23; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Tinnitus, Subjective; Tinnitus; Chronic Tinnitus
Keywords: Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Intervention Model Description: 2×2 factorial randomised controlled trial with two between-subjects factors: stimulation condition (real vs sham NITESGON) and listening condition (active auditory discrimination training vs passive listening during a visual task). Participants are assigned 1:1:1:1 to four parallel arms.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are blinded to stimulation condition (real vs sham NITESGON). Outcome assessors and data analysts are blinded to group allocation. The investigator operating the stimulation device does not take part in outcome assessments and follows coded procedures to deliver real or sham stimulation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Real Stimulation + Active Listening (ADT) (Experimental): Real stimulation delivered during active auditory frequency discrimination training.
  Interventions: Device: Real NITESGON; Behavioral: Active Listening
- Real Stimulation + Passive Listening (Active Comparator): Real stimulation delivered while participants perform a visual distractor task and are instructed to ignore auditory stimuli.
  Interventions: Device: Real NITESGON; Behavioral: Passive Listening (Control)
- Sham Stimulation + Active Listening (ADT) (Sham Comparator): Sham stimulation delivered during active auditory frequency discrimination training.
  Interventions: Device: Sham NITESGON; Behavioral: Active Listening
- Sham Stimulation + Passive Listening (Sham Comparator): Sham stimulation delivered while participants perform a visual distractor task and are instructed to ignore auditory stimuli.
  Interventions: Device: Sham NITESGON; Behavioral: Passive Listening (Control)

INTERVENTIONS:
Device: Real NITESGON — Real NITESGON is delivered transcutaneously via two saline-soaked sponge electrodes (35 cm² each) positioned bilaterally over the C2 dermatomes to target the greater occipital nerve. Stimulation consists of a 20 Hz sinusoidal current at 1.5 mA peak-to-peak, ramped up over 30 seconds and ramped down over 5 seconds. It is administered concurrently with the task for ~45 minutes per session, across eight sessions (2/week) over 4 weeks.
  Arms: Real Stimulation + Active Listening (ADT); Real Stimulation + Passive Listening
Device: Sham NITESGON — Sham NITESGON is delivered using two saline-soaked sponge electrodes (35 cm² each) positioned bilaterally over the C2 dermatomes. The sham condition mimics real stimulation sensations via a 30-second ramp-up followed by a brief ramp-down, with no sustained current thereafter. Sham is administered concurrently with the task for ~45 minutes per session, across eight sessions (2/week) over 4 weeks.
  Arms: Sham Stimulation + Active Listening (ADT); Sham Stimulation + Passive Listening
Behavioral: Active Listening — ADT is delivered using a three-interval, three-alternative forced-choice (3I-3AFC) frequency discrimination task. Standard tone frequencies are individually selected using ERB/critical-band spacing, centered one octave below each participant's dominant tinnitus pitch and extending to lower frequencies; the highest standard is kept below the tinnitus pitch region. Tones are presented binaurally via headphones, with presentation levels calibrated to individual audiometric thresholds and matched for equal SPL in both ears.
  Other Names: Auditory frequency discrimination training (ADT)
  Arms: Real Stimulation + Active Listening (ADT); Sham Stimulation + Active Listening (ADT)
Behavioral: Passive Listening (Control) — VisDT uses a three-interval, three-alternative forced-choice (3I-3AFC) paradigm with Gabor patches (sinusoidal gratings windowed by a Gaussian envelope) of fixed spatial frequency (6 cycles/degree) and fixed spatial spread; on each trial, one interval contains an orientation deviant relative to the standard. During VisDT, participants attend to the visual task while concurrent binaural tones are presented passively using a predetermined, non-adaptive schedule. Auditory tones are individually calibrated to audiometric thresholds and drawn from ERB-spaced frequencies centered one octave below the dominant tinnitus pitch and extending to lower frequencies, with the highest frequency kept below the tinnitus pitch region.
  Other Names: Visual distractor task (VisDT)
  Arms: Real Stimulation + Passive Listening; Sham Stimulation + Passive Listening

SUMMARY:
This study tests whether pairing non-invasive stimulation of the greater occipital nerve (NITESGON) with an attentionally demanding auditory frequency discrimination training task reduces tinnitus loudness and tinnitus-related distress. One hundred adults with chronic tonal tinnitus will be randomised to one of four groups in a 2×2 factorial design: real versus sham NITESGON and active versus passive listening during auditory stimulation. Participants complete eight sessions across four weeks, with outcomes assessed at baseline, end of treatment, 28 days post-treatment, and 6 months post-treatment.

DETAILED DESCRIPTION:
This is a single-centre, prospective, double-blind, placebo-controlled, 2×2 factorial randomised controlled trial conducted at Trinity College Dublin. The intervention combines transcutaneous electrical stimulation targeting the greater occipital nerve (NITESGON) with auditory stimulation delivered during a structured training paradigm. The two between-subjects factors are stimulation condition (real NITESGON vs sham NITESGON) and listening condition (active listening: auditory frequency discrimination training vs passive listening: visual distractor task while auditory stimuli are presented). One hundred adults with chronic tonal tinnitus will be randomised 1:1:1:1 to one of four arms. Participants complete eight sessions (two per week for four weeks). Primary outcomes-tinnitus loudness (VAS 0-100), tinnitus-related functional impact (TFI 0-100), and tinnitus handicap (THI 0-100)-and secondary outcomes are assessed at baseline (T0), end of treatment (T1), 28 days after treatment completion (T2), and 6 months after treatment completion (T3). Secondary outcomes include tinnitus psychoacoustics, extended high-frequency audiometry, speech-in-noise performance, EEG (resting-state and auditory oddball), autonomic/biomarker measures (pupillometry, heart rate, saliva), patient global impression of change, quality of life, and safety/blinding assessments.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-80 years
* Continuous subjective tinnitus for >3 months and ≤5 years
* Predominantly tonal tinnitus (unilateral or bilateral)
* Screening THI score 28-76
* Minimum Masking Level (MML) 20-80 dB HL
* No prior tinnitus neuromodulation treatment
* Able to comply with eight sessions over four weeks and follow-up assessments

Exclusion Criteria:

* Objective tinnitus or predominantly somatic tinnitus
* Pulsatile tinnitus
* Evidence of conductive hearing loss (abnormal otoscopy or tympanometry)
* Pure-tone audiometry exclusions: >40 dB HL at any frequency 250 Hz-1 kHz OR >80 dB HL at any frequency 2-8 kHz in either ear
* Hearing aid use initiated within the past 90 days
* Active implantable medical device (e.g., pacemaker, DBS, cochlear implant)
* LDL <30 dB SL at 500 Hz in either ear
* Diagnosis of temporomandibular joint disorder or occipital neuralgia
* Severe anxiety (STAI >120/160)
* Cognitive impairment (MMSE <25)
* Severe depressive symptoms (BDI ≥30)
* Diagnosis of Menière's disease
* Current pregnancy
* Involvement in medicolegal cases
* History of auditory hallucinations
* Current prescription of central nervous system drugs likely to alter neuromodulatory function (e.g., noradrenergic, dopaminergic, serotonergic, benzodiazepine, cholinergic, or other psychoactive medications)
* Currently enrolled in another interventional study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2029-01-30 (Estimated)

PRIMARY OUTCOMES:
Tinnitus Loudness (Visual Analogue Scale, VAS 0-100) | Baseline visit, end of treatment at 4 weeks, 28 days post-treatment, and 6 months post-treatment.
  0-100 mm VAS anchored from "not audible" to "extremely loud"; higher scores indicate greater perceived tinnitus loudness.
Tinnitus Functional Index (TFI, 0-100) | Baseline visit, end of treatment at 4 weeks, 28 days post-treatment, and 6 months post-treatment.
  25-item self-report measure of tinnitus-related functional impact; total score 0-100, higher scores indicate greater impairment.
Tinnitus Handicap Inventory (THI, 0-100) | Baseline visit, end of treatment at 4 weeks, 28 days post-treatment, and 6 months post-treatment.
  25-item measure of tinnitus-related handicap; total score 0-100, higher scores indicate greater handicap.

SECONDARY OUTCOMES:
Audiometry (Extended High-Frequency Thresholds up to 13 kHz) | Baseline visit, end of treatment at 4 weeks, 28 days post-treatment, and 6 months post-treatment.
  Air-conduction pure-tone audiometry thresholds will be measured from 250 Hz up to 13 kHz (extended high-frequency audiometry) to characterise hearing status and support calibration of stimulus sensation levels.
Speech-in-Noise Performance (e.g., QuickSIN) | Baseline visit, end of treatment at 4 weeks, 28 days post-treatment, and 6 months post-treatment.
  Speech perception in noise will be assessed using a standardised speech-in-noise test administered in a controlled environment.
Patient Global Impression of Change (PGIC) | End of treatment at 4 weeks, 28 days post-treatment, and 6 months post-treatment.
  Participant-rated global change since baseline using the Patient Global Impression of Change (PGIC) scale (-3 = very much worse to +3 = very much improved; higher scores indicate greater improvement).
Quality of Life (World Health Organization Quality of Life-BREF questionnaire) | Baseline visit, end of treatment at 4 weeks, 28 days post-treatment, and 6 months post-treatment.
  Quality of life assessed using the World Health Organization Quality of Life-BREF (WHOQOL-BREF), yielding domain scores and an overall score (0-100; higher scores indicate better quality of life).
Adverse Events (Stimulation Side-Effects Questionnaire) | Up to 4 weeks (Sessions 1-8)
  Stimulation tolerability assessed each visit using a Stimulation Side-Effects Questionnaire recording presence and severity of side effects (e.g., tingling, itching, headache) rated on a numeric severity scale (0-10; higher scores indicate worse side effects), plus event frequency.
Tinnitus Pitch Matching | Baseline, end of treatment at 4 weeks, 28 days post-treatment, and 6 months post-treatment.
  Dominant tinnitus pitch estimated by psychoacoustic pitch matching and recorded as frequency in hertz (Hz).
Tinnitus Loudness Matching and Discomfort Levels | Baseline visit, end of treatment at 4 weeks, 28 days post-treatment, and 6 months post-treatment.
  Loudness matching and discomfort levels: Tinnitus loudness matching recorded in decibels sensation level (dB SL; dB above audiometric threshold) at the matched frequency, and loudness discomfort levels recorded in decibels sensation level (dB SL; dB above threshold) at tested frequencies.
Minimum Masking Level (MML) | Baseline visit, end of treatment at 4 weeks, 28 days post-treatment, and 6 months post-treatment.
  Broadband noise level required to fully mask tinnitus, recorded in decibels hearing level (dB HL).
Resting-State EEG Spectral Power (Eyes Closed) | Baseline visit, end of treatment (4 weeks), 28 days post-treatment, and 6 months post-treatment.
  Resting-state eyes-closed electroencephalography (EEG) spectral power averaged within prespecified frequency bands and electrode/network regions, reported in decibels (dB); higher values indicate greater spectral power.
Resting-State EEG Functional Connectivity (Eyes Closed) | Baseline visit, end of treatment (4 weeks), 28 days post-treatment, and 6 months post-treatment.
  Resting-state eyes-closed EEG functional connectivity within prespecified networks, quantified as phase-locking value (PLV; unitless, 0-1); higher values indicate stronger phase synchronization.
Auditory Oddball Task-Evoked Response Amplitude | Baseline visit, end of treatment (4 weeks), 28 days post-treatment, and 6 months post-treatment.
  Auditory oddball event-related potential (ERP) amplitude (e.g., P300) averaged over prespecified electrodes/time windows, reported in microvolts (µV); higher absolute amplitude indicates larger task-evoked response.
Auditory Oddball Task-Evoked Response Latency | Baseline visit, end of treatment (4 weeks), 28 days post-treatment, and 6 months post-treatment.
  Auditory oddball ERP component latency (e.g., P300 peak latency) within prespecified time windows, reported in milliseconds (ms); lower values indicate faster evoked responses.
Pupillometry | Baseline visit, end of treatment (4 weeks), 28 days post-treatment, and 6 months post-treatment.
  Task-related pupil diameter during pupillometry, summarized as mean (or peak) pupil size change from baseline, reported in millimeters (mm); larger values indicate greater pupil dilation.
Heart Rate | Baseline visit, end of treatment (4 weeks), 28 days post-treatment, and 6 months post-treatment.
  Electrocardiography (ECG)-derived heart rate, reported in beats per minute (bpm); higher values indicate faster heart rate.
Saliva Biomarkers | Baseline visit, end of treatment (4 weeks), 28 days post-treatment, and 6 months post-treatment.
  Concentration of prespecified salivary biomarkers of arousal/neuromodulatory engagement, reported in nanograms per milliliter (ng/mL) (or assay-specific units); higher values indicate higher biomarker concentration.

CONTACTS AND LOCATIONS:
Locations (1):
- Trinity College Institute of Neuroscience (TCIN), Dublin, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Undecided